CLINICAL TRIAL: NCT03543800
Title: Comparison of Conventional Platelet-Rich Plasma Treatment of Osteoarthritic Knee With a New Autologous Blood Product (CytoRich)
Brief Title: PRP Treatment of Osteoarthritic Knee With a New Autologous Blood Product (CytoRich)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Antnor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GA-777
Record Dates: First submitted 2018-05-22; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABP (Experimental): (test treatment)
  Interventions: Device: Cytorich PRP kit
- PRP (Active Comparator): (active control)
  Interventions: Device: PRP kit

INTERVENTIONS:
Device: Cytorich PRP kit — Subjects randomized to the PRP treatment arm will receive PRP only without the anti-inflammatory component of ABP added
  Arms: ABP
Device: PRP kit — PRP kit legally marketed in Canada for PRP
  Arms: PRP

SUMMARY:
This study is aimed at evaluating the efficacy and safety of Cytorich compared to platelet-rich plasma (PRP) in alleviating pain and improving function in subjects with knee OA.

DETAILED DESCRIPTION:
This active-controlled, randomized, double-blind, prospective study will enroll subjects with knee OA. Subjects will be randomized equally to treatment with 4 injections of ABP (test treatment) or 4 injections of PRP (active control).

ELIGIBILITY:
Inclusion Criteria:

* Radiographic confirmation of OA in the knee and screening knee pain score of >50 mm on a 100 mm visual analog scale (VAS) for at least one knee.

Exclusion Criteria:

* Female who is pregnant, lactating, or unwilling to use adequate contraception during the clinical study.
* Subject who had viscosupplementation within 3 months of screening.
* Subject treated with non-steroidal anti-inflammatory drugs (NSAIDs) within 72 hours of screening.
* Subject who received steroid treatment within 8 weeks of screening.
* Subject who had an acute disease or trauma within 6 weeks of screening.
* Subject with any major surgery, arthoplasty or arthroscopy in the target knee or lower extremities within 6 weeks of screening (or any planned surgeries throughout the duration of the study).
* Subject with a major dysplasia or congenital abnormality of the knee or a condition which may affect the knee (i.e., osteonecrosis, chondrocalcinosis).
* Subject with a primary inflammatory arthropathy (i.e., rheumatoid arthritis, psoriatic arthritis, gouty arthritis).
* Subject with knee joint infection, skin diseases, or infections in or near the area of injection.
* Subject with any musculoskeletal condition that would impede measurement of the effectiveness at the knee (in particular symptomatic hip OA).
* Subject with any claudication or peripheral vascular disease.
* Subject with active malignancy or that has been in treatment for a malignancy within the past 3 years.
* Subject with uncontrolled diabetes mellitus, diabetic neuropathy, or complications from infection.
* Subject with known sensitivity to citric acid.
* Subject taking oral or parental anticoagulant therapy other than acetylsalicylic acid 325 mg per day or less.
* Subject with active disease that may require periodic treatment with systemic steroids during the study period.
* Subject with other diseases or conditions as assessed by the Investigator that may limit the ability to perform necessary study evaluations (e.g., active alcohol abuse, active drug abuse, significant psychiatric or neurological disorders, planned relocation, etc.) or any other factors (e.g., ongoing litigation for workers compensation for musculoskeletal injuries or disorders) that may compromise the subject's ability to participate in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-02-04 (Actual); Primary Completion 2019-05-20 (Estimated); Study Completion 2019-05-20 (Estimated)

PRIMARY OUTCOMES:
VAS pain score | Week 12 (Day 85) compared to baseline for ABP and PRP
  Change in VAS pain score

SECONDARY OUTCOMES:
WOMAC pain and function score | Week 12 (Day 85) compared to baseline for ABP and PRP
  Change in WOMAC pain and function score

CONTACTS AND LOCATIONS:
Overall Officials: Ira Brokhman, PhD, Study Director — Galea Clinic
Locations (1):
- Galea Clinic, Etobicoke, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided